CLINICAL TRIAL: NCT06027203
Title: Freehand Transperineal Prostate Biopsies Without Antibiotic Prophylaxis - the New Gold Standard?
Brief Title: Transperineal Versus Transrectal Prostate Biopsy
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MUMC-Pbx23
Record Dates: First submitted 2023-07-18; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
Keywords: prostate biopsy; prostate cancer; transperineal; transrectal
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- transrectal biopsy
  Interventions: Procedure: prostate biopsy
- transperineal biopsy
  Interventions: Procedure: prostate biopsy

INTERVENTIONS:
Procedure: prostate biopsy — Prostate biopsy by either transrectal or transperineal technique

SUMMARY:
Background: Prostate biopsies are essential to diagnose prostate cancer (PCa). Transrectal prostate biopsies (TR-PB) are commonly performed, however disadvantages include the requirement of antibiotic prophylaxis (AP) and higher complication rates than transperineal prostate biopsies (TP-PB). Guidelines still recommend the use of AP for TP-PB due to the limited evidence regarding complication rates after their omission. However, the rising rates of antibiotic resistance is of concern. The aim of this study was to compare the complication and detection rates of freehand TP-PB without AP versus TR-PB with AP.

Methods: This single center retrospective study was performed in an academic hospital. TP-PB were introduced in 2019 and implemented as the main technique by late 2020. To compare the two techniques, data was collected for freehand TR-PB with AP between 2017-2018 and freehand TP-PB without AP between 2021-2022. The data from 2019 and 2020 were excluded to rule out the effects of the initial learning curve during the transition period. Primary outcome measure was post-biopsy complications occurring within 2 weeks, focusing on infectious complications. Secondary outcome measures were detection rates and upgrading/reclassification in the repeat biopsy in active surveillance (AS). Statistical analysis was performed using a Fisher exact or Chi-Squared test.

ELIGIBILITY:
Inclusion Criteria:

* men who underwent prostate biopsy between 2017-2018 (transrectal)
* men who underwent prostate biopsy between 2012-2022 (transperineal)

Exclusion Criteria:

* positive urine culture before biopsy
* patients in the transrectal biopsy group who did not take the prescribed course of antibiotic prophylaxis
* incomplete medical dossier where the occurrence of a complication could not be assessed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All men who underwent a transrectal prostate biopsy between January 2017 and December 2018, and/or a transperineal prostate biopsy between January 2021 and December 2022 in the Urology department of MUMC+
Sampling Method: Non-Probability Sample
Enrollment: 923 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Complications | 2 weeks
  Urinary tract infections, urinary retention, hematuria

SECONDARY OUTCOMES:
Detection rate | 2 weeks
  Chance of detecting prostate cancer according to histopathology of needle biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided